CLINICAL TRIAL: NCT03542032
Title: Comparison of I -Gel Mask Airway Placement Methods in Elective Surgery: Jaw Thrust Maneuver vs Conventional Technique
Brief Title: Comparison of I-Gel Laryngeal Mask Airway Placement Methods in Elective Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Diskapi Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ilkay baran akkuş, principle investigator, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: I-Gel
Record Dates: First submitted 2018-05-18; First posted 2018-05-31 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2018-05

CONDITIONS: Effective I -Gel Mask Airway Placement Technique
Keywords: i-gel; jaw-thrust

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- jaw-thrust (Other): the i-gel was inserted with triple airway maneuver (mouth opening, head extension and jaw thrust) This groups will record the insertion time of i-gel, number of trials, operative time, placement complications.
  Recorded complications (blood, laryngospasm, etc.) during insertion and removal of supraglottic airway devices will be assessed.
  Patients' postoperative sore throat will be questioned and recorded.
  Interventions: Other: i-gel placement maneuvers
- classic group (No Intervention): In the classic group, the index finger used as a guide, pushes the back of i-gel towards the hard palate, inserting it into the pharynx till a resistance is felt and the i-gel is then fixed it its place. This groups will record the insertion time of i-gel, number of trials, operative time, placement complications.
  Recorded complications (blood, laryngospasm, etc.) during insertion and removal of supraglottic airway devices will be assessed.
  Patients' postoperative sore throat will be questioned and recorded.

INTERVENTIONS:
Other: i-gel placement maneuvers — the i-gel was inserted with triple airway maneuver (mouth opening, head extension and jaw thrust) In the classic maneuver , the index finger used as a guide, pushes the back of i-gel towards the hard palate, inserting it into the pharynx till a resistance is felt and the i-gel is then fixed it its place.
  Arms: jaw-thrust

SUMMARY:
To compare the jaw thrust maneuver with the conventional technical methods to place the I-Gel laryngeal mask

DETAILED DESCRIPTION:
Patients who underwent elective surgery under general anesthesia and who were between the ages of 18 and 75 and who had ASA score I-II-III would be included in the study. Patients' mallampati scores, thyromental distances, mouth openings will be recorded.

Patients will be divided into two groups according to supraglottic airway insertion method.

Both groups will record the insertion time of i-gel, number of trials, operative time, placement complications.

Recorded complications (blood, laryngospasm, etc.) during insertion and removal of supraglottic airway devices will be assessed.

Patients' postoperative sore throat will be questioned and recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 18 and 75 years
2. American Society of Anesthesiologists I, II or III

Exclusion Criteria:

1. Those with anatomical disorders related to the upper airway
2. lung disease
3. gastric regurgitation
4. Those who have had lung infection in the last 3 weeks
5. Supraglottic airway vehicle not settled
6. Those who are hired for any reason
7. EtCO2> 45

American Society of Anesthesiologists 4 or 5

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
insertion time | 2 minutes
  Time for successful i-gel insertion
successful insertion number | 2 minutes
  successful insertion number

CONTACTS AND LOCATIONS:
Locations (1):
- Diskapi Yildirim Beyazit Training Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No